CLINICAL TRIAL: NCT04593446
Title: Difference of Surgical Site Infection Between Using Sodium Picosulfate Solution(PicosolutionⓇ) and Oral Sulfate Tablet(ORA·FANGⓇ) in Colorectal Cancer Surgery : Phase II. Prospective, Randomised, Multicenter, Non-inferiority Trial
Brief Title: Difference of Surgical Site Infection Between Using Sodium Picosulfate Solution(PicosolutionⓇ) and Oral Sulfate Tablet(ORA·FANGⓇ) in Colorectal Cancer Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: Seoul National University Hospital (Other); Seoul National University Bundang Hospital (Other); Daehang Hospital (Other)
Responsible Party: Principal Investigator, Sung Sil Park, Clinical Professor, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC2020-0138
Record Dates: First submitted 2020-10-12; First posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Colorectal Cancer
Keywords: sodium picosulfate solution; oral sulfate tablet; surgical site infection
MeSH Terms: conditions — Colorectal Neoplasms; Surgical Wound Infection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Sulfate Tablet(ORA·FANGⓇ) (Experimental): Subjects who are randomized into experimental arm will receive 14 pills at 8 pm in the evening 2days before the surgery and another 14 pills on 6am in the morning 1day before the surgery
  Interventions: Drug: Oral Sulfate Tablet(ORA·FANGⓇ)
- Sodium Picosulfate Solution(PicosolutionⓇ) (Active Comparator): Subjects who are randomized into experimental arm will receive 170ml of solution with at 8 pm in the evening 2days before the surgery and another 170ml of solution on 6am in the morning 1day before the surgery
  Interventions: Drug: Sodium Picosulfate Solution(PicosolutionⓇ)

INTERVENTIONS:
Drug: Oral Sulfate Tablet(ORA·FANGⓇ) — Subjects who are randomized into experimental arm will receive 14 pills at 8 pm in the evening 2days before the surgery and another 14 pills on 6am in the morning 1day before the surgery
  Subjects who are randomized into comparator will receive 170ml of solution with at 8 pm in the evening 2days before the surgery and another 170ml of solution on 6am in the morning 1day before the surgery
  Arms: Oral Sulfate Tablet(ORA·FANGⓇ)
Drug: Sodium Picosulfate Solution(PicosolutionⓇ) — Sodium Picosulfate Solution(PicosolutionⓇ)
  Arms: Sodium Picosulfate Solution(PicosolutionⓇ)

SUMMARY:
This is a prospective randomized study to evaluate the difference in the rate of surgical site infection between the patients who used Sodium Picosulfate solution(PicosolutionⓇ) and tablet Oral Sulphate Solution(ORA·FANGⓇ) for bowel preparation before colorectal cancer surgery .

DETAILED DESCRIPTION:
It has been reported that tablet oral sulphate solution(ORA·FANGⓇ) showed a successful bowel cleansing rate of 95.5%, which is similar to compared to sodium picosulfate solution(PicosolutionⓇ).

In terms of the rate of surgical site infection(SSI), sodium picosulfate solution(PicosolutionⓇ) showed 8% of SSI rate. However there is no report for the SSI rate of tablet oral sulphate solution(ORA·FANGⓇ). We aimed to compare the SSI rates between these two group.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are scheduled for an elective minimally invasive surgery for colorectal cancer
2. ASA score, 2 or less

Exclusion Criteria:

1. Bowel obstruction
2. FAP or IBD patients
3. Emergency operation
4. Pregnancy
5. Breast feeding
6. Severe medical condition such as severe cardiac,hepatic, or renal failure (creatinine ≥ 3.0 mg/dL (normal 0.8-1.4 mg/dL)),
7. Allergy to drug and refusal to participate in the study

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 414 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
The rate of surgical site infection | 30 days
  The operator will evaluate the rate of the surgical site infection during the postoperative hospitalization period or the first outpatient visit after surgery. We will use the definition of surgical site infection published in 1999 by the Centers for Disease Control and Prevention (CDC).

SECONDARY OUTCOMES:
The quality of the bowel preparation | during surgery
  The operator will evaluate he quality of the bowel preparation using Arohchick bowel preparation scale during the surgery.
  Aronchick scale Excellent:5, good:4, fair:3, poor:2, inadequate:1
The patient's tolerability for bowel preparation | 1 day after bowel preparation
  Using questionnaire, the tolerance will be scored after bowel preparation
  Tolerability score Very comfortable: 5 Comfortable: 4 Fair: 3 Uncomfortable: 2 Very uncomfortable: 1

CONTACTS AND LOCATIONS:
Overall Officials: Hyoung-Chul Park, Doctor, Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center, Korea, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No